CLINICAL TRIAL: NCT03869710
Title: Analgesic Effects of Ultrasound-guided Dry-Needling Therapy for Neck and Head Pain by Active and Latent Myofascial Trigger Points.
Brief Title: Analgesic Effects of Ultrasound-guided Dry-Needling Therapy for Neck and Head Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of COVID pandemic
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Principal Investigator, San Salvatore Hospital of L'Aquila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0209913/17
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Neck Pain; Head Pain
Keywords: Pain
MeSH Terms: conditions — Neck Pain; Headache; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dry-Needling (Experimental): Ultrasound-Guided Dry-Needling Therapy focused on the active and latent myofascial trigger points.
  Interventions: Device: Ultrasound-guided Dry-Needling Therapy

INTERVENTIONS:
Device: Ultrasound-guided Dry-Needling Therapy — The needle will be insert under ultrasound guidance to elicit the myofascial response on the neck of the patients

SUMMARY:
The analgesic effects of ultrasound-guided dry-needling therapy will be evaluated in the management of head and neck pain.

DETAILED DESCRIPTION:
The analgesic effects of ultrasound-guided dry-needling therapy will be evaluated in the management of head and neck pain by myofascial active and latent trigger point.

The myofascial pain control will be assessed for the superficial and deep posterolateral muscle complex of neck. The analgesic request, Range Of Motion (ROM), Motion Related Pain (MRP) and the quality of life, will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain
* Chronic head pain

Exclusion Criteria:

* previous surgery of neck and head
* Body Mass Index > 39,99
* politrauma patients
* pregnancy
* neck and head infections

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-12-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Trigger Point | The first hour of the treatment
  The number of the elicited myofascial trigger points assessed during dry-needling treatment

SECONDARY OUTCOMES:
Analgesic request | 3 months trom treatment
  The analgesic request will be assessed in mg of equianalgesic morphine
Karnofsky Performance Status | 3 months from treatment
  The quality of life assessed by Karnofsky Performance Status (a 0-100 steps scale, from 0 [Dead] to 100 [Normal no complaints; no evidence of disease]).
Range Of Motion (ROM) | 3 months after treatment
  The alpha angle expressed in degrees and assessed during
Motion Related Pain | 3 months after treatment
  Pain assessed by Numeric Rating Scale (a 10-steps scale, from 0 [no pain] to 10 [worse pain]), during flexion, extension and rotation of neck and head
Perception | 3 months after treatment
  Pain assessed by Numeric Rating Scale (a 10-steps scale, from 0 [no pain] to 10 [worse pain])

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Fusco, MD, Principal Investigator — San Salvatore Academic Hospital
Locations (1):
- San Salvatore Academic Hospital, Coppito, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No